CLINICAL TRIAL: NCT02091869
Title: A Randomized Trial Examining the Effectiveness of Mobile-Based Asthma Action Plans vs. Paper Asthma Action Plans
Acronym: PEAK2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202623
Record Dates: First submitted 2014-01-14; First posted 2014-03-19 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: Adolescents; Asthma; Asthma Symptoms
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paper Asthma Action Plan (Experimental): Participants will utilize a paper-based asthma action plan to record asthma symptoms, peak flows, and medication usage.
  Interventions: Other: Paper Asthma Action Plan
- Mobile Phone (Experimental): Participants will record asthma symptoms, medication usage, and peak flow data on their phones.
  Interventions: Device: Mobile Phone

INTERVENTIONS:
Other: Paper Asthma Action Plan — Participants will utilize a paper based asthma action plan to record asthma symptoms and medication usage.
  Arms: Paper Asthma Action Plan
Device: Mobile Phone — Participant will be able to log peak flow data, medications, and symptoms in their mobile phones utilizing the mobile app.
  Other Names: IPhone and Android mobile phones
  Arms: Mobile Phone

SUMMARY:
The purpose of this study is to see if using a mobile phone application asthma action plan will help improve asthma management.

DETAILED DESCRIPTION:
The investigators propose to conduct a randomized trial to examine the effectiveness of a mobile-based Asthma Action Plan that will meet the national guidelines recommendation for individualized Asthma Action Plan treatment plans. The mobile app will provide immediate instructions and feedback once data is entered by the participants. This is an randomized trial which will be compared with an paper asthma action plan. Participants will be randomized through a statistical table. The mobile app will be password and Health Information Portability and Protection Act protected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and ≤ 17 years.
* Access to Apple or Android based smart phone
* Mild to severe persistent asthma or poorly controlled asthma (see definitions below).

  o A different assessment of eligibility will be performed depending on whether or not the parent reports use of a preventive asthma medication at baseline. This is consistent with 2007 National Asthma Education Prevention Program recommendations that make a strong distinction between classifying asthma severity (for children not using preventive medications) and assessing control (for children using preventive medications). If a child has used a preventive medication in the past, but reports no use of the medication in the prior 3 months, we will assess severity.)
* Children not using a preventive medication at baseline: Assess for mild persistent to severe persistent asthma. Any 1 of the following, during the prior 4 weeks (as defined by parent interview in the waiting room) will determine severity:

  * An average of >2 days per week with asthma symptoms
  * >2 days per week with rescue medication use
  * ≥2 nights per month awakened with nighttime symptoms
  * Minor limitation of activity
  * ≥2 episodes of asthma during the past year that have required systemic corticosteroids
* Children using a preventive medication at baseline: Assess for poorly controlled asthma. Any 1 of the following, during the prior 4 weeks (as defined by parent interview in the waiting room) will determine control:

  * An average of >2 days per week with asthma symptoms
  * >2 days per week with rescue medication use
  * ≥2 nights per month awakened with nighttime symptoms
  * Some limitation of activity
  * ≥2 episodes of asthma during the past year that have required systemic corticosteroids.

Exclusion Criteria:

* Significant underlying respiratory disease other than asthma (such as cystic fibrosis or chronic lung disease) that could potentially interfere with asthma-related outcome measures.
* Significant co-morbid conditions (such as moderate to severe developmental delay, i.e. special education classroom or diagnosis) that could preclude participation in an education-based intervention.
* Inability to speak or understand English (child or parent).
* Children in foster care or other situations in which consent cannot be obtained from a guardian.
* Prior enrollment in the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T Perry, MD,FAAP, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Moorman JE, Rudd RA, Johnson CA, King M, Minor P, Bailey C, Scalia MR, Akinbami LJ; Centers for Disease Control and Prevention (CDC). National surveillance for asthma--United States, 1980-2004. MMWR Surveill Summ. 2007 Oct 19;56(8):1-54. PMID 17947969
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Forero R, Bauman A, Young L, Larkin P. Asthma prevalence and management in Australian adolescents: results from three community surveys. J Adolesc Health. 1992 Dec;13(8):707-12. doi: 10.1016/1054-139x(92)90068-m. PMID 1290773
- [Background] Kyngas HA. Compliance of adolescents with asthma. Nurs Health Sci. 1999 Sep;1(3):195-202. doi: 10.1046/j.1442-2018.1999.00025.x. PMID 10894643
- [Background] Braun-Fahrlander C, Gassner M, Grize L, Minder CE, Varonier HS, Vuille JC, Wuthrich B, Sennhauser FH. Comparison of responses to an asthma symptom questionnaire (ISAAC core questions) completed by adolescents and their parents. SCARPOL-Team. Swiss Study on Childhood Allergy and Respiratory Symptoms with respect to Air Pollution. Pediatr Pulmonol. 1998 Mar;25(3):159-66. doi: 10.1002/(sici)1099-0496(199803)25:33.0.co;2-h. PMID 9556007
- [Background] Venn A, Lewis S, Cooper M, Hill J, Britton J. Questionnaire study of effect of sex and age on the prevalence of wheeze and asthma in adolescence. BMJ. 1998 Jun 27;316(7149):1945-6. doi: 10.1136/bmj.316.7149.1945. No abstract available. PMID 9641931
- [Background] Calmes D, Leake BD, Carlisle DM. Adverse asthma outcomes among children hospitalized with asthma in California. Pediatrics. 1998 May;101(5):845-50. doi: 10.1542/peds.101.5.845. PMID 9565412
- [Derived] Perry TT, Marshall A, Berlinski A, Rettiganti M, Brown RH, Randle SM, Luo C, Bian J. Smartphone-based vs paper-based asthma action plans for adolescents. Ann Allergy Asthma Immunol. 2017 Mar;118(3):298-303. doi: 10.1016/j.anai.2016.11.028. Epub 2017 Jan 19. PMID 28111110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paper Asthma Action Plan | Mobile Phone
Started | 17 | 17
Completed | 17 | 14
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paper Asthma Action Plan | Mobile Phone | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 17 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 15.4 [13.4 to 16.1] | 15.3 [14.4 to 16.8] | 15.4 [14.5 to 16.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Test Scores
Description: The Asthma Control Test™ (ACT) is a 5 question health survey used to measure asthma control in individuals 12 years of age and older. The total sum scores range from 5-25. Higher scores mean that asthma is more controlled. The ACT is an efficient, reliable, and valid method of measuring asthma control, with or without, lung functioning measures such as spirometry. ACT helps identify and detect asthma patients who are not well controlled. ACT scores were examined pre- and post-intervention. A score total of 19 or less means asthma may not be well controlled. The timeframe is during the past 4 weeks. The scale range for Question 1 is "all the time" (1) to "none of the time" (5); Question 2 range: "more than once a day" (1) to "not at all" (5); Question 3 range: "4 or more nights a week" (1) to "not at all" (5); Question 4 range: "3 or more times per day" (1) to "not at all" (5); Question 5 range: "not controlled at all" (1) to "completely controlled" (5).
Time Frame: Baseline and Six months
Population: Our staff biostatistician used a random number generator using ANCOVA model to assign all participants into either the mobile app or paper app groups per protocol. The biostatistician was not be involved in testing or intervention procedures.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Paper Asthma Action Plan | Mobile Phone
Number analyzed (Participants) | 17 | 17
units on a scale
  Six Months, All Participants | 21 [17 to 22] | 22 [21 to 24]
  Baseline, All Participants | 20 [17 to 24] | 21 [18 to 24]

2. Secondary Outcome: Change in Asthma Self-Efficacy Scores
Description: The Child Self-Efficacy instrument is a 14 item validated questionnaire designed to measure the child's self-efficacy with regard to attack prevention and attack management. The child will be required to select one of 5 responses ranging from "not at all sure" (1 point); "a little bit sure" (2 points); "fairly sure" (3 points); "quite sure" (4 points) to "completely sure" (5 points). Total score range from 14-70. The attack prevention scale range from 6-30 and attack management range from 8-40. The higher score represent a greater degree of self-efficacy. The Cronbach's α reliability = 0.75. The child self-efficacy questionnaire will be administered at baseline (pre-intervention) and at the end of the intervention (post-intervention).
Time Frame: Baseline and Six months
Population: Our staff biostatistician used a random number generator using ANCOVA model to assign all participants into either the mobile app or paper app groups per protocol.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Paper Asthma Action Plan | Mobile Phone
Number analyzed (Participants) | 17 | 17
units on a scale
  6 Month (Prevention) Post Intervention | 36 [34 to 38] | 34 [32 to 37]
  Baseline (Prevention) | 35 [33 to 38] | 35 [34 to 37]
  6 Month (Management) Post Intervention | 25 [24 to 28] | 27 [24 to 28]
  Baseline (Management)) | 26 [22 to 28] | 25 [23 to 28]

3. Other Pre Specified Outcome: Comparison of Participant Usage Rates Between Mobile and Paper Asthma Action Plans
Description: We measured the participant usage rates by frequency of a mobile asthma action plan compared to usage rates of a paper asthma action plan. No mobile usage data was collected for the paper asthma plan group; and no paper usage data was collected for mobile phone group.
Time Frame: Six months
Population: Our staff biostatistician used a random number generator using ANCOVA model to assign all participants into either the mobile app or paper app groups per protocol. Three participants did not use the mobile app per protocol.
Measure: Median (Full Range); unit: days per week
Arm/Group | Paper Asthma Action Plan | Mobile Phone
Number analyzed (Participants) | 17 | 14
days per week
  Mobile Use (Average Days per Week) | NA [NA to NA] — This was not assessed in the paper asthma action plan group. | 4.36 [2.81 to 6.51]
  Paper Use (Average Days per Week) | 7.00 [6.97 to 7.00] | NA [NA to NA] — This was not assessed in the mobile phone group.

4. Other Pre Specified Outcome: Comparison of Participant Usage Rates Between Mobile and Paper Asthma Action Plans
Description: as for outcome 3
Time Frame: Six months
Population: Mobile phone usage was not assessed in the paper asthma action plan group.
Measure: Median (Full Range); unit: times per week
Arm/Group | Paper Asthma Action Plan | Mobile Phone
Number analyzed (Participants) | 0 | 17
times per week |  | 12.17 [7.16 to 16.46]

ADVERSE EVENTS:
Arm/Group | Paper Asthma Action Plan | Mobile Phone
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
There were not limitations and caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No